CLINICAL TRIAL: NCT03170245
Title: Adiponectin, Interleukin-6 (IL-6) and High Sensitive C-reactive Protein (hsC-RP) in Relation to Carotid Intima-media Thickness in B-thalassemia Patients
Brief Title: Adiponectin, IL-6 and hsC-RP in Relation to Carotid Intima-media Thickness in B-thalassemia Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Hussein, Principal investigator, Assiut University
Other Study IDs: ADICIBT
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Carotid Intima-Media Thickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and serum to be used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- B thalassemia group: Laboratory investigations :
  * complete blood count
  * renal and liver function tests
  * serum ferritin
  * lipid profile
  * Interleukin -6
  * HsC-RP
  * Adiponectin level
  Imaging :
  * Abdominal ultrasound
  * Echocardiography
  * Carotid intima media thickness
  Interventions: Diagnostic Test: Interleukin-6; Diagnostic Test: HsC-RP; Diagnostic Test: Adiponectin level; Diagnostic Test: Carotid intima media thickness
- Control group: Laboratory investigations :
  * complete blood count
  * renal and liver function tests
  * serum ferritin
  * lipid profile
  * Interleukin -6
  * HsC-RP
  * Adiponectin level
  Imaging :
  * Abdominal ultrasound
  * Echocardiography
  * Carotid intima media thickness
  Interventions: Diagnostic Test: Interleukin-6; Diagnostic Test: HsC-RP; Diagnostic Test: Adiponectin level; Diagnostic Test: Carotid intima media thickness

INTERVENTIONS:
Diagnostic Test: Interleukin-6 — serum samples used for doing the test by ELISA
Diagnostic Test: HsC-RP — serum samples used for doing the test by ELISA
Diagnostic Test: Adiponectin level — serum samples used for doing the test by ELISA
Diagnostic Test: Carotid intima media thickness — Done by carotid doppler

SUMMARY:
Every year, 100,000 neonates are born with hemoglobinopathies around the world. Thalassemia is the most common heterogeneous disease of the human being . It is a disease of high prevalence in Mediterranean, Indian, North Chinese, and Pacific populations. Recently, the quantity and quality of the life of these patients have been significantly improved by regular transfusion and iron chelating therapy .

DETAILED DESCRIPTION:
β-thalassemia result from a decrease in β- globin chains which result in a relative excess of α-globin chains . Approximately 1.5% of the population is estimated to be carriers for β-thalassemia . Around 60,000 new births are recorded to be affected by β-thalassemia per year in the world . In Egypt, it was estimated that 1000/1.5 million live births per year suffer from thalassemia; β -thalassemia is the most common type, with a carrier rate starting from 5.3%-9% . Depending on severity of hematological and clinical conditions, β-thalassemia is classified into three types, namely, β-thalassemia minor (β-TMI) (also called as carrier), β-thalassemia intermedia (β-TI) and β-thalassemia major (β-TM). The clinical severity of β-thalassemia intermedia has ranged from asymptomatic carrier state to severe transfusion-dependent type. β-Thalassemia minor is clinically asymptomatic but can be characterized by specific hematological features .

A high incidence of thromboembolic event has been observed in patients with β -thalassemia. Endothelial dysfunction occurred in those patients was attributed to peroxidative tissue injury because of continuous blood transfusions . Carotid atherosclerosis was positively associated with serum ferritin independent of traditional cardiovascular risk factors and transfusion-related iron overload in β-thalassemia major (β-TM) has been associated with the onset of cardiovascular complications, including cardiac dysfunction and vascular anomalies. Increased iron overload has also been reported in patients with non-transfusion dependent thalassemia (NTDT) Direct iron-related injury is responsible for different kinds of cardiovascular abnormalities, including progressive worsening of diastolic and systolic ventricular function, increased arterial stiffness and pulmonary hypertension .

It has previously demonstrated that both patients with β-TM and β-TI exhibit a global impairment of arterial vasorelaxation and increased carotid intima-media thickness (cIMT) as compared with control healthy subjects , those findings strongly support the notion that the severe arterial dysfunction in thalassemia may indicate an additional clinical vulnerability for venous thromboembolism. Epidemiologically, vascular events appear at a relatively young age with a four times higher incidence in β-TI as compared with β-TM patients . Carotid intima-media thickness is related both with incident and prevalent cardiovascular disease and is accepted measure of subclinical atherosclerosis . It also increases the risk for future myocardial infarction (MI) .

Lipid abnormalities have been detected in different types of β -thalassemia, and also in various hematological disorders including sickle cell disease, glucose-6-phosphate dehydrogenase (G6PD) deficiency, spherocytosis, aplastic anemia and myelodysplastic syndrome . Patients with β - thalassemia are at risk of developing premature atherosclerosis because of those abnormalities .

Inflammatory biomarkers including C-reactive proteins and cytokines (IL-6) are found to be increased in various inflammatory conditions and have been used by a number of workers as biomarker of inflammation in thalassemia . The iron laden insult to the tissues in transfusion dependent thalassemic patients has been monitored using the high sensitive C-reactive proteins as biomarker of inflammation and vascular risk .

High Sensitive C-reactive protein(hsC-RP)is clinically proven as a method to predict vascular risk and to enhance event rates in clinical trials. As hsC-RP and IL-6 levels measured in apparently healthy populations also predict future vascular risk; hsC-RP and IL-6 levels have been shown to correlate with endothelial dysfunction, arterial stiffness, and extent of subclinical atherosclerosis . IL-6 signaling has also been linked to plaque initiation and destabilization , to microvascular flow dysfunction , and to adverse outcomes in the setting of acute ischemia .

Adiponectin, an adipose tissue secreted protein, has been well recognized to exhibit insulin-sensitizing, anti-inflammatory and anti-atherosclerotic properties . Its level is associated with atherosclerosis markers such as inflammation, oxidative stress, and endothelial dysfunction . Its anti-inflammatory action, resulting in decreased production and inhibition of tumor necrosis factor-α (TNF-α) action, decreased IL-6 production, and human studies previously reported an inverse association between adiponectin level and C-RP , TNF-α and IL-6 .

Adiponectin varies according to body mass index with lower levels in obese individuals , in type 2 diabetes mellitus (T2DM) and in hypertensive patients.

Circulating low adiponectin levels (hypoadiponectinemia) is considered an independent risk factor for endothelial dysfunction and modulating vessel wall health . It has been correlated with elevated risk factors of atherosclerotic cardiovascular disease and associated with hypertension, dyslipidemia, and inflammation in both the general population and in diabetic patients .

ELIGIBILITY:
Inclusion Criteria:

* B thalassemia patients

Exclusion Criteria:

* Diabetes mellitus
* Hypertension
* Obesity

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All B thalassemia parients who admitted to Clinical Hematology Unit - Internal Medicine Department at Assiut University Gospital
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Adiponectin | once (1 day)
  Estimated by ElISA

SECONDARY OUTCOMES:
HsC-reactive protein | once (1 day)
  By ELISA
Interleukin-6 | once (1 day)
  By ELISA
carotid intima media thickness | once (1 day)
  By carotid doppler

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahalis G, Kremastinos DT, Terzis G, Kalogeropoulos AP, Chrysanthopoulou A, Karakantza M, Kourakli A, Adamopoulos S, Tselepis AD, Grapsas N, Siablis D, Zoumbos NC, Alexopoulos D. Global vasomotor dysfunction and accelerated vascular aging in beta-thalassemia major. Atherosclerosis. 2008 Jun;198(2):448-57. doi: 10.1016/j.atherosclerosis.2007.09.030. Epub 2007 Nov 7. PMID 17988670
- [Background] Stoyanova E, Trudel M, Felfly H, Lemsaddek W, Garcia D, Cloutier G. Vascular endothelial dysfunction in beta-thalassemia occurs despite increased eNOS expression and preserved vascular smooth muscle cell reactivity to NO. PLoS One. 2012;7(6):e38089. doi: 10.1371/journal.pone.0038089. Epub 2012 Jun 19. PMID 22723848
- [Background] Hahalis G, Kalogeropoulos A, Terzis G, Tselepis AD, Kourakli A, Mylona P, Grapsas N, Alexopoulos D. Premature atherosclerosis in non-transfusion-dependent beta-thalassemia intermedia. Cardiology. 2011;118(3):159-63. doi: 10.1159/000327997. Epub 2011 Jun 1. PMID 21646780
- [Background] Chen YG, Lin CL, Ho CL, Chen YC, Kao CH. Risk of coronary artery disease in transfusion-naive thalassemia populations: A nationwide population-based retrospective cohort study. Eur J Intern Med. 2015 May;26(4):250-4. doi: 10.1016/j.ejim.2015.02.001. Epub 2015 Feb 18. PMID 25704855
- [Background] Tantawy AA, Adly AA, El Maaty MG, Amin SA. Subclinical atherosclerosis in young beta-thalassemia major patients. Hemoglobin. 2009;33(6):463-74. doi: 10.3109/03630260903343616. PMID 19958191
- [Background] Lee WY, Allison MA, Kim DJ, Song CH, Barrett-Connor E. Association of interleukin-6 and C-reactive protein with subclinical carotid atherosclerosis (the Rancho Bernardo Study). Am J Cardiol. 2007 Jan 1;99(1):99-102. doi: 10.1016/j.amjcard.2006.07.070. Epub 2006 Nov 9. PMID 17196470
- [Background] Guo F, Dong M, Ren F, Zhang C, Li J, Tao Z, Yang J, Li G. Association between local interleukin-6 levels and slow flow/microvascular dysfunction. J Thromb Thrombolysis. 2014 May;37(4):475-82. doi: 10.1007/s11239-013-0974-0. PMID 24242026
- [Background] Prakash J, Mittal B, Awasthi S, Srivastava N. Association of adiponectin gene polymorphism with adiponectin levels and risk for insulin resistance syndrome. Int J Prev Med. 2015 Apr 8;6:31. doi: 10.4103/2008-7802.154773. eCollection 2015. PMID 25949781
- [Background] Kriketos AD, Greenfield JR, Peake PW, Furler SM, Denyer GS, Charlesworth JA, Campbell LV. Inflammation, insulin resistance, and adiposity: a study of first-degree relatives of type 2 diabetic subjects. Diabetes Care. 2004 Aug;27(8):2033-40. doi: 10.2337/diacare.27.8.2033. PMID 15277436
- [Background] Kim DH, Kim C, Ding EL, Townsend MK, Lipsitz LA. Adiponectin levels and the risk of hypertension: a systematic review and meta-analysis. Hypertension. 2013 Jul;62(1):27-32. doi: 10.1161/HYPERTENSIONAHA.113.01453. Epub 2013 May 28. PMID 23716587
- [Background] Okui H, Hamasaki S, Ishida S, Kataoka T, Orihara K, Fukudome T, Ogawa M, Oketani N, Saihara K, Shinsato T, Shirasawa T, Mizoguchi E, Kubozono T, Ichiki H, Ninomiya Y, Matsushita T, Nakasaki M, Tei C. Adiponectin is a better predictor of endothelial function of the coronary artery than HOMA-R, body mass index, immunoreactive insulin, or triglycerides. Int J Cardiol. 2008 May 7;126(1):53-61. doi: 10.1016/j.ijcard.2007.03.116. Epub 2007 May 2. PMID 17477992
- [Background] Attar MJ, Mohammadi S, Karimi M, Hosseinnezhad A, Hosseini SH, Eshraghian MR, Jafari N, Rahmani M, Karimi F, Nezhad MK. Association of adiponectin with dietary factors and cardiovascular risk factors in type 2 diabetes mellitus patients. Diabetes Metab Syndr. 2013 Jan-Mar;7(1):3-7. doi: 10.1016/j.dsx.2013.02.027. Epub 2013 Mar 9. PMID 23517787
- [Derived] Ahmad Ibrahim O, Ahmad AB, Nigm DA, Hussien AN, Mohammad Ibrahim WH. Subclinical atherosclerotic predictive value of inflammatory markers in thalassemia intermedia patients. Expert Rev Hematol. 2021 Jul;14(7):669-677. doi: 10.1080/17474086.2021.1959316. Epub 2021 Aug 6. PMID 34296962